CLINICAL TRIAL: NCT06846983
Title: Peripheral Perfusion Index As an Early Predictor of Successful Caudal Block in Pediatric Patients Undergoing Lower Abdominopelvic Surgeries Under General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD325/2024
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Perfusion Index; Caudal Block
Keywords: Peripheral perfusion index; caudal block; predictor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Peripheral perfusion index pulse oximeter — Masimo pulse oximeter probe for measuring peripheral perfusion index and predicting success of caudal block
  Other Names: Masimo pulse oximeter

SUMMARY:
The aim of this study is to assess early predictability of peripheral perfusion index to success of caudal block in pediatric patients undergoing lower abdominopelvic surgeries

DETAILED DESCRIPTION:
The aim of this study is to assess early predictability of peripheral perfusion index to success of caudal block in pediatric patients undergoing lower abdominopelvic surgeries. Preoperative assessment will be done which includes full history taking, clinical examination, standard laboratory investigations. Demographic data (age, weight, and sex) will be recorded.

All patients will be instructed to fast for 6 hours preoperatively while allowing clear fluids up to 2 hours prior to anesthesia as per the standard nil per oral (NPO) guidelines.

In the operating room, all patients will be monitored during the operation using: electrocardiography (ECG), pulse oximeter (SpO2), automated non-invasive arterial pressure (NIAP) measurement cuff, end tidal carbon dioxide (capnogram), volatile anesthetic monitoring, core temperature monitoring using a nasopharyngeal probe, and Masimo pulse oximeter probe for measuring PPI which will be applied to the big toe of the patient's foot and wrapped with gauze to reduce heat loss and to avoid the interference of ambient light.

Normothermia will be maintained using warm intravenous fluids and a forced air warm blanket.

Induction of general anesthesia will be done using inhalational sevoflurane at 8%, and after loss of consciousness, a peripheral intravenous access will be placed under complete aseptic condition. Fentanyl citrate at 1 µg/kg will be slowly injected intravenously then laryngeal mask with appropriate size will be inserted.

Maintenance of anesthesia will be with 50% oxygen-air mixture, and sevoflurane titrated to a minimum alveolar concentration MAC of 2%. Ringer acetate will be administered as the intraoperative maintenance fluid at the rate of 6 mL/kg/h.

The baseline value of PPI, heart rate (HR), and mean arterial pressure (MAP) will be recorded, corresponding to the value at 0 minute (T0) measured after induction of general anesthesia and before caudal block in supine position. The caudal block will be performed under complete aseptic conditions with the patient in the left lateral decubitus position with the hips and knees flexed using the landmark technique. Sterilization by Povidone Iodine will take place and insertion of the cannula will begin till appreciating the loss of resistance at which the needle is will be held and the cannula is advanced. After negative aspiration for blood and cerebrospinal fluid, 1mL/kg of 0.25% of bupivacaine hydrochloride will be injected at the rate of 1mL/3s and the patient will be turned supine immediately and surgical skin incision will be allowed to start 10 minutes after.

Following the caudal block, PPI, HR, and MAP will be recorded at 2, 5, 7, 10 (at skin incision), 15, and 20 minutes. Successful caudal block will be predicted as any or both of the following criteria achieved, whichever occurred earlier:

* ≥100% increase of PPI value from baseline.
* No tachycardia or hypertension on surgical stimulation (HR or MAP increase > 20% of baseline).

Percentage of successful blocks predicted with these criteria will be plotted against postoperative pain score as a main determinant of caudal block success with successful block defined as the following:

• Postoperative pain score as assessed by Children and Infants' Postoperative Pain Scale (CHIPPS) at 0 h and 30 min postoperatively is <4 out of 10.

A failed caudal block is defined based on failure to achieve the aforementioned criteria. And in case of block failure, an intravenous bolus of 1-2 ug/kg fentanyl will be administered intraoperatively, and a rescue post-operative analgesia in the form of bolus intravenous nalbuphine at a dose of 0.2 mg/kg will be provided to patients accordingly.

Patients will be divided into two groups based on success of the block: group (S) caudal success group, and group (F) caudal failure group. Both groups will receive the standard management (caudal block under general anesthesia) for the required procedure. There will not be a control group for this study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aging between 1-5 years of both sexes.
* Pediatric patients posted for elective lower abdominopelvic surgeries under general anesthesia (duration of surgery under 120 minutes).
* ASA physical status classes I - II.

Exclusion Criteria:

* Guardian's refusal of procedure or participation in the study.
* ASA classes III or above.
* Infection at site of injection.
* Neurological diseases and disorders such as (neuromuscular disease, cerebral palsy, spinal dysraphism …etc.)
* Coagulopathy and bleeding disorders.
* Hypersensitivity to the study medications.
* Patients receiving vasoactive drugs or beta blockers.
* Patients undergoing emergency surgery.
* Patients in active clinical sepsis.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients undergoing elective lower abdominopelvic surgeries under general anesthesia at El-Demerdash Pediatric Surgery Hospital during the study period. Surgeries include inguinal / inguinoscrotal hernia repair, hydrocelectomy, orchiopexy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
peripheral perfusion index predictability | From enrollment to discharge from post anesthesia care unit
  Monitor and compare peripheral perfusion index values before and after administration of the caudal block to determine if there is a significant correlation between early PPI changes and the success of caudal block

CONTACTS AND LOCATIONS:
Overall Officials: Omar Mohamed Taha Abdallah El-Safty, M.B.B.CH., MD., Study Chair — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data might not provide further insight to research work. yet, if found helpful to further studies planned IPD sharing will be considered

REFERENCES:
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Zielinski J, Morawska-Kochman M, Zatonski T. Pain assessment and management in children in the postoperative period: A review of the most commonly used postoperative pain assessment tools, new diagnostic methods and the latest guidelines for postoperative pain therapy in children. Adv Clin Exp Med. 2020 Mar;29(3):365-374. doi: 10.17219/acem/112600. PMID 32129952
- [Background] Wolf AR. Effects of regional analgesia on stress responses to pediatric surgery. Paediatr Anaesth. 2012 Jan;22(1):19-24. doi: 10.1111/j.1460-9592.2011.03714.x. Epub 2011 Oct 14. PMID 21999144
- [Background] Wiegele M, Marhofer P, Lonnqvist PA. Caudal epidural blocks in paediatric patients: a review and practical considerations. Br J Anaesth. 2019 Apr;122(4):509-517. doi: 10.1016/j.bja.2018.11.030. Epub 2019 Feb 1. PMID 30857607
- [Background] Toyama S, Kakumoto M, Morioka M, Matsuoka K, Omatsu H, Tagaito Y, Numai T, Shimoyama M. Perfusion index derived from a pulse oximeter can predict the incidence of hypotension during spinal anaesthesia for Caesarean delivery. Br J Anaesth. 2013 Aug;111(2):235-41. doi: 10.1093/bja/aet058. Epub 2013 Mar 21. PMID 23518802
- [Background] Szostek AS, Saunier C, Elsensohn MH, Boucher P, Merquiol F, Gerst A, Portefaix A, Chassard D, De Queiroz Siqueira M. Effective dose of ephedrine for treatment of hypotension after induction of general anaesthesia in neonates and infants less than 6 months of age: a multicentre randomised, controlled, open label, dose escalation trial. Br J Anaesth. 2023 May;130(5):603-610. doi: 10.1016/j.bja.2022.12.006. Epub 2023 Jan 12. PMID 36639328
- [Background] Suresh S, Ecoffey C, Bosenberg A, Lonnqvist PA, de Oliveira GS Jr, de Leon Casasola O, de Andres J, Ivani G. The European Society of Regional Anaesthesia and Pain Therapy/American Society of Regional Anesthesia and Pain Medicine Recommendations on Local Anesthetics and Adjuvants Dosage in Pediatric Regional Anesthesia. Reg Anesth Pain Med. 2018 Feb;43(2):211-216. doi: 10.1097/AAP.0000000000000702. PMID 29319604
- [Background] Sun X, He H, Xu M, Long Y. Peripheral perfusion index of pulse oximetry in adult patients: a narrative review. Eur J Med Res. 2024 Sep 11;29(1):457. doi: 10.1186/s40001-024-02048-3. PMID 39261939
- [Background] Silvani P, Camporesi A, Agostino MR, Salvo I. Caudal anesthesia in pediatrics: an update. Minerva Anestesiol. 2006 Jun;72(6):453-9. PMID 16682915
- [Background] Sekimoto K, Tobe M, Saito S. Local anesthetic toxicity: acute and chronic management. Acute Med Surg. 2017 Mar 6;4(2):152-160. doi: 10.1002/ams2.265. eCollection 2017 Apr. PMID 29123854
- [Background] Rajan K, Dave N, Dias R, Muneshwar P, Kesarkar N, Saxena V. Perfusion index as a predictor of working pediatric caudal block under general anesthesia- A prospective observational study. J Anaesthesiol Clin Pharmacol. 2022 Oct-Dec;38(4):635-639. doi: 10.4103/joacp.JOACP_34_21. Epub 2022 Dec 26. PMID 36778797
- [Background] Piasek CZ, Van Bel F, Sola A. Perfusion index in newborn infants: a noninvasive tool for neonatal monitoring. Acta Paediatr. 2014 May;103(5):468-73. doi: 10.1111/apa.12574. Epub 2014 Feb 23. PMID 24471645
- [Background] Nemeth M, Miller C, Brauer A. Perioperative Hypothermia in Children. Int J Environ Res Public Health. 2021 Jul 15;18(14):7541. doi: 10.3390/ijerph18147541. PMID 34299991
- [Background] Menzies R, Congreve K, Herodes V, Berg S, Mason DG. A survey of pediatric caudal extradural anesthesia practice. Paediatr Anaesth. 2009 Sep;19(9):829-36. doi: 10.1111/j.1460-9592.2009.03116.x. PMID 19691690
- [Background] Kubica-Cielinska A, Zielinska M. The use of nalbuphine in paediatric anaesthesia. Anaesthesiol Intensive Ther. 2015;47(3):252-6. doi: 10.5603/AIT.2015.0036. PMID 26165241
- [Background] • Elfeil YE, Zarad AR, Deghidy EA. Comparison of two different methods as reliable predictors of successful caudal block in children. Egypt J Anaesth. 2024; 40(1): 69-74.
- [Background] • El-Sonbaty M, El-Sonbaty A. Evaluation of Perfusion index (PI) efficiency in pediatric caudal block: Is it the time to depend on PI? Med J Cairo Univ. 2015; 83:223-7.
- [Background] Coutrot M, Dudoignon E, Joachim J, Gayat E, Vallee F, Depret F. Perfusion index: Physical principles, physiological meanings and clinical implications in anaesthesia and critical care. Anaesth Crit Care Pain Med. 2021 Dec;40(6):100964. doi: 10.1016/j.accpm.2021.100964. Epub 2021 Oct 24. PMID 34687923
- [Background] Benka AU, Pandurov M, Galambos IF, Rakic G, Vrsajkov V, Draskovic B. [Effects of caudal block in pediatric surgical patients: a randomized clinical trial]. Braz J Anesthesiol. 2020 Mar-Apr;70(2):97-103. doi: 10.1016/j.bjan.2019.12.003. Epub 2020 Feb 20. PMID 32204919
- [Background] Baduni N, Sanwal MK, Vajifdar H, Agarwala R. Postoperative analgesia in children: A comparison of three different doses of caudal epidural morphine. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):220-3. doi: 10.4103/0970-9185.182106. PMID 27275053
- [Background] Allen J. Photoplethysmography and its application in clinical physiological measurement. Physiol Meas. 2007 Mar;28(3):R1-39. doi: 10.1088/0967-3334/28/3/R01. Epub 2007 Feb 20. PMID 17322588